CLINICAL TRIAL: NCT04044482
Title: Evaluation of Health Related Quality of Life and Patient Adherence in Case of Hungarian Patients Affected by Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Other Study IDs: 24950-3/2016/EKU
Record Dates: First submitted 2019-07-24; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Translation and Cross-cultural adaptation process of the Osteoarthritis Knee and Hip Quality of Life questionnaire. According to granted guidelines, shared by the developer of the questionnaire, the study was conducted among Hungarian patients affected by osteoarthrosis.

DETAILED DESCRIPTION:
This prospective study was performed among patients diagnosed - by the doctors acting as the expert panel of this study - with OA of the lower limb. The recruitment period was: June 2017 and November 2017, in six hospitals situated in six different geographical regions of Hungary. The participating hospitals were selected in a way to represent different geographic and cultural areas of the country; the patients were selected randomly by the doctors of the given sites. The process was conducted with the contribution of: (1) Translation committee (4 members), (2) Our research team, as moderator (4 members), (3) Expert panel (6 doctors professors of the study sites: orthopaedists, rheumatologists, musculoskeletal rehabilitation doctors). The used instruments were for the validation process: Short version of World Health Organization Quality of life questionnaire (WHOQoL-BREF), EuroQuality of Life - 5-dimension questionnaire as generic quality of life measurement tools (EQ-5D - VAS). In addiction 99 patients filled the questionnaires in an appropriate way. The results were evaluated by 23.0 version of SPSS program.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* clinically/doctor diagnosed knee and/or hip osteoarthritis
* native Hungarian language
* ability of self-filling and completely filled patient data sheet.

Exclusion Criteria:

* age under 18 years
* other type of OA osteoarthritis
* psychiatric disorders
* surgeries within 1 month
* incapable of filling out the forms/tools

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both sex, above 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Validity and Reliability of the translated and adapated questionnaire | 17 months
  The translated questionnaire was tested among affected patients. First of all the face and content validity were evaluated, namely how understandable is the translated questionnaire for patients with Hungarian native language. How many percent of the items were no answered. According to the shared guideline if more then 5 % of an item is not answered should be selected from the final version of the questionnaire - with the exception of the items based on sexual life(3 items). The research team noticed that face and content validity were adequate.